CLINICAL TRIAL: NCT03525080
Title: Diagnostic Assessment Study, Single Site and Prospective, comparing18F-DOPA PET and Multiparametric RMI in Initial Exploration of Diffuse Glial Tumors
Brief Title: Comparison of 6-fluoro-[18F]-L-dihydroxyphenylalanine (18F-DOPA) Positron Emission Tomography (PET) and Multiparametric Resonance Magnetic Imagery (RMI) in Initial Exploration of Glial Tumors
Acronym: GLIROPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center Eugene Marquis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-4-52-010
Record Dates: First submitted 2018-05-02; First posted 2018-05-15 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Brain Neoplasms; Adult Brain Tumor
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET Arm (Experimental)
  Interventions: Diagnostic Test: PET imagery

INTERVENTIONS:
Diagnostic Test: PET imagery — Every patients will have a PET imagery in addition to standard MRI

SUMMARY:
For patient having a brain tumor, RMI is the standard exam for tumor characterization and determines initial surgery.

The aim of this study is to assess if PET could provide additional information that could have an impact on surgery (indication and planification)

ELIGIBILITY:
Inclusion Criteria:

* Suspected glial resectable tumor
* Free and informed consent
* Affiliated to French social security

Exclusion Criteria:

* Suspected high grade glioma
* Surgical emergency
* Pregnant or breastfeeding woman
* Patient deprived of their liberty or under guardianship
* Patient not able to follow study medical monitoring for geographical, social or psychological reasons
* Treated with carbidopa, catechol-O-methyl transferase inhibitor, haloperidol, reserpine within 2 weeks before PET imagery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2019-09-11 (Actual)

PRIMARY OUTCOMES:
PET pictures and MRI sequences comparison | Imagings performed up to 29 days after inclusion (before brain surgery)
  Comparison of PET pictures and MRI sequences will be done in order to assess concordance between both imagings

CONTACTS AND LOCATIONS:
Overall Officials: Florence LE JEUNE, Professor, Principal Investigator — Centre Eugène Marquis
Locations (1):
- Centre Eugène Marquis, Rennes, Brittany Region, France